CLINICAL TRIAL: NCT04855682
Title: EuroPainClinicsStudy X (Minimally Invasive Spinal Surgical Approaches)
Brief Title: EuroPainClinicsStudy X
Acronym: EPCS X
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Europainclinics z.ú. (Other)
Collaborators: R-CLINIC s.r.o. (Other); Faculty Hospital Nitra (Other); Slovak Academy of Sciences (Other Government); University Hospital Bratislava (Other)
Responsible Party: Principal Investigator, MUDr. Miroslav Buriánek MBA, MUDr. Robert Rapčan FIPP, Clinical Research Manager, R-CLINIC s.r.o.
Other Study IDs: 4184/2021/ODDZ-11156
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Endoscopic discectomy
  Interventions: Other: Retrospective observation after 24 months after the spinal procedure; Other: Retrospective observation after 12 months after the spinal procedure; Other: Prospective evaluation of patients after 12 and 24 months after the spinal procedure
- B: Microdisectomy
  Interventions: Other: Retrospective observation after 24 months after the spinal procedure; Other: Retrospective observation after 12 months after the spinal procedure; Other: Prospective evaluation of patients after 12 and 24 months after the spinal procedure
- C: Hemilaminectomy
  Interventions: Other: Retrospective observation after 24 months after the spinal procedure; Other: Retrospective observation after 12 months after the spinal procedure; Other: Prospective evaluation of patients after 12 and 24 months after the spinal procedure

INTERVENTIONS:
Other: Retrospective observation after 24 months after the spinal procedure — Retrospective evaluation of patients before the procedure, and prospective evaluation of patients 24 months after the spinal procedure, comparing the MRI changes and procedure impact on fatty muscle degeneration process
  Other Names: Quality of life; MRI description
Other: Retrospective observation after 12 months after the spinal procedure — Retrospective evaluation of the patient status before the procedure, and prospective evaluation of patients for 12 months after the spinal procedure, comparing the MRI changes
  Other Names: Quality of life; MRI description
Other: Prospective evaluation of patients after 12 and 24 months after the spinal procedure — Prospective evaluation of patients after 12 and 24 months after the spinal procedure, comparing the MRI changes
  Other Names: Quality of life; MRI description

SUMMARY:
Non-interventional, retrospective-prospective cohort study based on the collection of data and their evaluation after medical procedures: micro-discectomy, endoscopic discectomy, and hemilaminectomy.

DETAILED DESCRIPTION:
The aim of this clinical study is to compare the benefits and complications after minimally invasive spinal procedures in patients with acute lumbosacral radicular syndrome caused by a herniated disc compressing the spinal neural structures.

The study only works with patient data provided by the outpatient clinic for research analysis in the EPCS IV clinical study. All patient data are encrypted during collection and evaluation during the study, and stored in an encrypted database. The data will be evaluated by an independent institution - The Institute of Measurement of the Slovak Academy of Sciences.

ELIGIBILITY:
Inclusion Criteria:

* patient age 18-60 years
* first spinal surgery in the areas L1-S1
* signed informed consent for the participation in the study

Exclusion Criteria:

* patients with a history of other back problems (compression fracture, spondylitis, tumour)
* patients after repeated spinal surgeries
* patients with a systemic disease affecting the muscles elite athletes
* patients who disagree to participate in the study
* women with a positive pregnancy test or women planning on becoming pregnant

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after medical procedures: micro-discectomy, endoscopic discectomy, and hemilaminectomy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Fat degeneration of muscles | 12 months after procedure
  Fat degeneration of musculus erector spinae and multifidus muscles evaluated by comparing the pre-operative current MRI of the lumbosacral spine using the 2-point Dixon Technique and Goutallier classification in each group
Fat degeneration of muscles | 24 months after procedure
  Fat degeneration of musculus erector spinae and multifidus muscles evaluated by comparing the pre-operative current MRI of the lumbosacral spine using the 2-point Dixon Technique and Goutallier classification in each group
Oswestry disability index (ODI) | 12 months and 24 months after procedure
  ODI is based on a questionnaire, which includes 10 items, each one has 6 possible answers. Each item is rated from 0 to 5 and the sum of all answers is evaluated on a scale from 0-100, with higher scores meaning more serious symptoms.
Oswestry disability index (ODI) | 24 months after procedure
  ODI is based on a questionnaire, which includes 10 items, each one has 6 possible answers. Each item is rated from 0 to 5 and the sum of all answers is evaluated on a scale from 0-100, with higher scores meaning more serious symptoms.
EQ-5D-5L | 12 months after procedure
  EQ-5D is a standardized questionnaire tool developed by the EuroQol group as a measure of the quality of life linked to health, that can be used in a wide spectrum of health conditions and their treatment. The system has 5 dimensions: mobility, being able to take care of oneself, every-day activities, pain/discomfort and anxiety/depression. Each system can be graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems. T Changes in the visual analogue scale (VAS) of lower limb pain evaluated on a scale of 0 to 10
EQ-5D-5L | 24 months after procedure
  EQ-5D is a standardized questionnaire tool developed by the EuroQol group as a measure of the quality of life linked to health, that can be used in a wide spectrum of health conditions and their treatment. The system has 5 dimensions: mobility, being able to take care of oneself, every-day activities, pain/discomfort and anxiety/depression. Each system can be graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems. T Changes in the visual analogue scale (VAS) of lower limb pain evaluated on a scale of 0 to 10

SECONDARY OUTCOMES:
Usage of painkillers before and after the procedures | 12 months after procedure
Usage of painkillers before and after the procedures | 24 months after procedure
Occurrence of early and late post-surgery complications | 12 months after procedure
Occurrence of early and late post-surgery complications | 24 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Burianek, MD MBA, Study Chair — clinical monitor
Locations (1):
- R - Clinic s.r.o., Bardejov, Slovakia